CLINICAL TRIAL: NCT02053792
Title: A Phase 3b Open-label, Multicenter, Safety and Efficacy Extension Study of a Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) in Subjects With Hemophilia B
Brief Title: A Safety and Efficacy Extension Study of a Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Patients With Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL654_3003; 2012-005489-37 (EudraCT Number)
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — albutrepenonacog alfa

ARMS (1):
- rIX-FP (Experimental): Subjects will administer rIX-FP by intravenous infusion as routine prophylaxis, prevention, and on-demand treatment during a treatment period of approximately 3 years.
  The routine prophylaxis treatment interval for previously treated patients may be changed at each scheduled 6-month follow-up assessment. On-demand treatment with rIX-FP will be used for all bleeding episodes requiring treatment. Subjects (other than those in France) may participate in a surgical 'substudy' in which rIX-FP may be administered before, during and after surgery. An additional substudy will examine the safety and PK of subcutaneous administration of rIX-FP.
  For previously untreated patients, subjects will administer rIX-FP intravenously as weekly prophylaxis and/or on-demand treatment during the first 12 months, and as weekly routine prophylaxis thereafter.
  The dose of rIX-FP administered will be based on the subject's previous rIX-FP use and/or pharmacokinetic data.
  Interventions: Biological: rIX-FP

INTERVENTIONS:
Biological: rIX-FP — Recombinant Fusion Protein Linking Coagulation Factor IX with Albumin (rIX-FP)

SUMMARY:
This study will examine the long-term safety and efficacy of rIX-FP for the control and prevention of bleeding episodes in children and adults with severe hemophilia B. The study will include subjects who have not previously been treated with Factor IX products, subjects who previously completed a CSL-sponsored rIX-FP lead-in study and subjects requiring major non-emergency surgery who have not previously completed a CSL-sponsored rIX-FP lead-in study.

A surgical prophylaxis substudy will examine the efficacy of rIX-FP in subjects with hemophilia B who are undergoing non-emergency major or minor surgery. An additional substudy will examine the safety and PK of subcutaneous (SC) administration of rIX-FP.

ELIGIBILITY:
Inclusion criteria:

Main study inclusion criteria:

For previously treated subjects, either:

* Completed a CSL-sponsored rIX-FP (CSL654) study, including study CSL654_3001 [NCT01496274] or study CSL654_3002 [NCT01662531].

Or:

* Scheduled to have a major non-emergency surgery within approximately 8 weeks from the anticipated date of receiving the first rIX-FP injection.
* Not previously completed a CSL-sponsored rIX-FP lead-in study.
* Male, 12 to 70 years of age.
* Documented severe hemophilia B (FIX activity of ≤ 2%), or confirmed at screening by the central laboratory.
* Subjects who have received FIX products (plasma-derived and / or recombinant FIX) for > 150 exposure days (EDs), confirmed by their treating physician.
* No confirmed history of FIX inhibitor formation at screening by the central laboratory

For previously untreated subjects:

* Male, up to 18 years of age.
* Documented severe hemophilia B (FIX activity of ≤ 2%), or confirmed at screening by the central laboratory.
* Never previously been treated with FIX clotting factor products (except previous exposure to blood components).
* No confirmed history of FIX inhibitor formation

Surgery substudy inclusion criterion:

* Must require non-emergency surgery

Subcutaneous substudy inclusion criteria:

* Male, at least 18 years of age.
* Subjects currently enrolled in Study CSL654_3003
* Subjects who have received rIX-FP for ≥ 100 EDs (single-dose cohorts) or for ≥ 50 EDs (repeated-dose cohort)

Exclusion criteria:

Main study exclusion criteria:

* Currently receiving a therapy not permitted during the study.
* Any issue that, in the opinion of the investigator, would render the subject unsuitable for participation in the study.

For subjects who have previously completed a CSL-sponsored rIX-FP study:

* Unwilling to participate in the study for a total of 100 exposure days.

For subjects requiring major non-emergency surgery who have not previously completed a CSL-sponsored rIX-FP lead-in study:

* Known hypersensitivity (ie, allergic reaction or anaphylaxis) to any FIX product or hamster protein.
* Known congenital or acquired coagulation disorder other than congenital FIX deficiency.
* Currently receiving IV immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment.
* Low platelet count, kidney or liver disease.
* Human immunodeficiency virus positive with a CD4 count < 200/mm3.

For previously untreated subjects:

* Known congenital or acquired coagulation disorder other than congenital FIX deficiency (except for vitamin K deficiency of the newborn).
* Known kidney or liver dysfunction or any condition which, in the investigator's opinion, place the patient at unjustifiable risk.

The surgical substudy does not have any additional exclusion criteria, although subject(s) in France will not be eligible for the surgery sub-study.

Subcutaneous substudy exclusion criteria:

* Intravenous use of rIX-FP within 14 days of subcutaneous administration of rIX-FP.
* Life-threatening bleeding episode or major surgery during the 3 months prior to substudy entry

Max Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (42):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Indiana Hemophilia & Thrombosis Center Inc., Indianapolis, Indiana
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - The Children's Hospital Westmead, Westmead, Victoria
- Austria (2):
  - Department of Pediatrics, Medical University of Vienna, Vienna
  - Medical University of Vienna, Vienna General Hospital, Vienna
- SHAT "Joan Pavel" ODD [Hemorrhagic Diathesis & Anemia], Sofia, Bulgaria
- McMaster University, Hamilton, Ontario, Canada
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni Nemocrice Ostrava, Ostrava-Poruba
  - Fakultni nemocnice v Motole, Prague
- France (5):
  - CHRU Hopital Morvan, Brest
  - Hopital Louis Pradel, Bron
  - Hopital Bicetre - Centre de Traitement del'Hemophilia, Le Kremlin-Bicêtre
  - Hopital d'Enfants La Timonepital, Marseille
  - Hopital Necker-Enfants Malades, Paris
- Germany (7):
  - Institut fur experimentelle Hamatologie, Bonn
  - Prof. Hess Kinderklinik, Bremen
  - CRC Coagulation Research Centre GmbH, Duisburg
  - Heinrich Heine University Dusseldorf, Düsseldorf
  - Universtatsklinikum Hamburg-Eppendorf, Hamburg
  - Werlhof-Institute for Haemostasis and Thrombosis, Hanover
  - Kurpfalzkrankenhaus Heidlerberg GmbH, Heidelberg
- Chaim Sheba Medical Center, Tel Aviv, Israel
- Italy (3):
  - IRCCS Ospedale Maggiore[Centro emofilia e Trobosi], Milan
  - UOS Gestione e Organizzazione Funzlone Hub Emofilia, Parma
  - Centro Malattie Emorragiche e Trombotiche Ospedale, Vicenza
- Japan (7):
  - Nara Medical University Hospital, Kashihara
  - University of Occupational and Environmental Health, Kitakyushu
  - Nagoya University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Tokyo Medical University Hospital, Tokyo
  - Ogikubo Hospital, Tokyo
  - St. Marianna University, School of Medicine, Seibu Hospital, Yokohama
- National Blood Center, Kuala Lumpur, Malaysia
- Perpetual Succour Hospital, Cebu, Philippines
- Haemophilia Comprehensive Care Centre, Parktown, South Africa
- Spain (3):
  - C.H.U. A Coruna, A Coruña
  - Hospital Vall Hebron, Barcelona
  - H.U. La Paz, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 115 male previously treated patients (PTPs) and previously untreated patients (PUPs) with hemophilia B were planned to be enrolled, including all eligible PTPs from CSLB-sponsored rIX-FP lead-in studies, approximately 10 PTPs who required major, nonemergency surgery, and approximately 20 PUPs.
Groups:
- CSL654 (PTPs): Previously treated patients (PTPs) will administer CSL654 (rIX-FP) by intravenous infusion as routine prophylaxis, prevention, and on-demand treatment during a treatment period of approximately 5 years or the time it takes to reach 100 exposure days (EDs). The dose of rIX-FP administered will be based on the subject's previous rIX-FP use and/or pharmacokinetic data.
- CSL654 (PUPs): Previously untreated patients (PUPs) will administer CSL654 (rIX-FP) by intravenous infusion as weekly prophylaxis and/or on-demand treatment during the first 12 months, and as weekly routine prophylaxis thereafter up to 3 years or the time it takes to achieve 50 EDs. The dose of rIX-FP administered will be based on the pharmacokinetic data.
Period: Overall Study
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Started | 83 | 14
Completed | 77 | 10
Not Completed | 6 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Development of High titer FIX inhibitor | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — The patient was not compliant to the study procedure | 1 | 0
Not completed — Patient reached minimum number of exposure days and was allowed to stop | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CSL654 (PTPs): Previously treated patients (PTPs) will administer CSL654 (rIX-FP) by intravenous infusion as routine prophylaxis, prevention, and on-demand treatment during a treatment period of approximately 5 years or the time it took to reach 100 exposure days (EDs). The dose of rIX-FP administered will be based on the subject's previous rIX-FP use and/or pharmacokinetic data.
- CSL654 (PUPs): Previously untreated patients (PUPs) administered CSL654 (rIX-FP) intravenously as weekly prophylaxis and/or on-demand treatment during the first 12 months, and as weekly routine prophylaxis thereafter up to 3 years or the time it takes to achieve 50 EDs. The dose of rIX-FP administered will be based on the subject's previous rIX-FP use and/or pharmacokinetic data.
- Total: Total of all reporting groups
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs) | Total
Number analyzed (Participants) | 83 | 14 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 14 | 44
  Between 18 and 65 years | 53 | 0 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety Population (SP) was used. It was pre-specified in the Statistical Analysis Plan to collect age data separately for PTPs and PUPs and to not calculate the age for the total overall population.
  years
    CSL654 (PTPs): number analyzed (Participants) | 83 | 0 | 83
    CSL654 (PTPs) | 27.7 (17.81) |  | 27.7 (17.81)
    CSL654 (PUPs): number analyzed (Participants) | 0 | 12 | 12
    CSL654 (PUPs) |  | 1.3 (3.11) | 1.3 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 83 | 14 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: SP was used
  Participants
    number analyzed (Participants) | 83 | 12 | 95
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 81 | 12 | 93
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: SP was used
  Participants
    number analyzed (Participants) | 83 | 12 | 95
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 12 | 1 | 13
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 0 | 3
    White | 68 | 10 | 78
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Czechia | 3 | 0 | 3
  United States | 2 | 4 | 6
  Japan | 9 | 0 | 9
  Philippines | 1 | 1 | 2
  Malaysia | 2 | 0 | 2
  Spain | 6 | 0 | 6
  Canada | 1 | 0 | 1
  Austria | 4 | 1 | 5
  Italy | 10 | 2 | 12
  South Africa | 2 | 0 | 2
  Israel | 15 | 0 | 15
  Bulgaria | 4 | 0 | 4
  Australia | 2 | 3 | 5
  France | 14 | 0 | 14
  Germany | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Who Developed Inhibitors Against Factor IX (FIX)
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs). For PUPs: up to 3 years or the time it takes to achieve 50 EDs.
Population: Safety Population (SP) consisted of all participants who received ≥ 1 dose of rIX-FP during this study
Measure: Count of Participants; unit: Participants
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 83 | 12
Participants | 0 | 1

2. Primary Outcome: Mean Incremental Recovery of a 50 IU/kg Dose of CSL654 in Previously Untreated Patients (PUPs)
Description: Incremental Recovery: The increase in plasma concentration per IU/kg of factor administered.
Time Frame: Approximately 30 minutes after infusion of CSL654
Population: Pharmacokinetic (PK) Population consisted of participants who received ≥ 1 dose of rIX-FP and had a sufficient number of analyzable PK blood samples (ie, ≥ 1 PK parameter calculated) for the PK assessment of rIX-FP. Participants were excluded from the analyses if an insufficient number of analyzable PK samples was obtained to permit the evaluation of ≥ 1 PK parameter. Only PUPs were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 0 | 8
(IU/dL)/(IU/kg)
  Uncorrected FIX Activity |  | 1.295 (0.3578)
  Baseline-corrected FIX Activity |  | 1.231 (0.3729)

3. Secondary Outcome: Total Annualized Bleeding Rate (ABR) by Prophylaxis Regimen in Previously Treated Patients (PTPs)
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: Efficacy Population (EP) consisted of all participants in the Safety Population (SP). Only PTPs were analyzed for this endpoint. Participants were assigned under multiple regimens during the study, but were counted only once in any given regimen group. Annualized Bleeding Rate was derived only for subjects who were on the given regimen for at least 12 weeks.
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Participant
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 83 | 0
Bleeds/Year/Participant
  7-Day Regimen: number analyzed (Participants) | 41 | 0
  7-Day Regimen | 2.89 (3.115) |
  10-Day Regimen: number analyzed (Participants) | 23 | 0
  10-Day Regimen | 2.72 (2.827) |
  14-Day Regimen: number analyzed (Participants) | 48 | 0
  14-Day Regimen | 2.72 (3.395) |
  21-Day Regimen: number analyzed (Participants) | 11 | 0
  21-Day Regimen | 1.19 (1.572) |

4. Secondary Outcome: Spontaneous ABR by Prophylaxis Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: EP. Only PTPs were analyzed for this endpoint. Participants may be assigned under multiple regimens during the study, but will be counted only once in any given regimen group. Annualized Bleeding Rate is derived only for subjects who are on the given regimen for at least 12 weeks.
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Participant
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 83 | 0
Bleeds/Year/Participant
  7-Day Regimen: number analyzed (Participants) | 41 | 0
  7-Day Regimen | 0.95 (1.672) |
  10-Day Regimen: number analyzed (Participants) | 23 | 0
  10-Day Regimen | 0.98 (1.689) |
  14-Day Regimen: number analyzed (Participants) | 48 | 0
  14-Day Regimen | 1.32 (2.205) |
  21-Day Regimen: number analyzed (Participants) | 11 | 0
  21-Day Regimen | 0.60 (1.408) |

5. Secondary Outcome: Average Amount of CSL654 (rIX-FP) Consumed Per Month Per Subject During Routine Prophylaxis Treatment.
Time Frame: as for outcome 1
Population: EP
Measure: Mean (Standard Deviation); unit: IU/kg per month
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 83 | 12
IU/kg per month | 181.8 (35.16) | 188.53 (24.096)

6. Secondary Outcome: Percentage of Participants With at Least One Treatment Emergent Adverse Event (TEAE) and the Percentage of Participants With at Least One CSL654-related TEAE
Time Frame: as for outcome 1
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 83 | 12
percentage of participants
  AEs | 89.2 | 91.7
  Related AEs | 2.4 | 16.7

7. Secondary Outcome: Number of Participants With Investigator's Overall Clinical Assessment of Hemostatic Efficacy for the Treatment of Major Bleeding Events With CSL654 in PUPs
Description: The investigator will rate the efficacy of the rIX-FP treatment based on a hemostatic efficacy four point rating scale of excellent, good, moderate, or poor/no response.
Time Frame: Up to 3 years or the time it takes to achieve 50 EDs
Population: EP. This endpoint was for PUPs only. No major bleeding events were reported. Therefore, no data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 0 | 12
Participants |  | 0

8. Secondary Outcome: Total ABR for On-demand Regimen vs. 14-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: EP. Only PTPs were analyzed for this endpoint. Participants may be assigned under multiple regimens during the study, but will be counted only once in any given regimen group. Number of participants analyzed are those who received at least 12 weeks of treatment in the respective regimen.
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 14 | 0
Bleeds/Year/Subject
  On-demand Regimen | 17.51 (7.130) |
  14-Day Regimen | 3.01 (4.204) |

9. Secondary Outcome: Spontaneous ABR for On-demand Regimen vs. 14-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 14 | 0
Bleeds/Year/Subject
  On-demand Regimen | 13.17 (5.873) |
  14-Day Regimen | 1.93 (3.363) |

10. Secondary Outcome: Total ABR for Subjects >=12 Years: 7-Day Regimen vs. 14-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 41 | 0
Bleeds/Year/Subject
  7-Day Regimen | 1.12 (1.697) |
  14-Day Regimen | 2.19 (3.000) |

11. Secondary Outcome: Spontaneous ABR for Subjects >=12 Years: 7-Day Regimen vs. 14-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 41 | 0
Bleeds/Year/Subject
  7-Day Regimen | 0.49 (1.135) |
  14-Day Regimen | 1.33 (2.349) |

12. Secondary Outcome: Total ABR for Subjects >=12 Years: 7-Day Regimen vs. (10 or 14)-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 49 | 0
Bleeds/Year/Subject
  7-Day Regimen | 1.31 (1.868) |
  (10 or 14)-Day Regimen | 2.01 (2.700) |

13. Secondary Outcome: Spontaneous ABR for Subjects >=12 Years: 7-Day Regimen vs. (10 or 14)-Day Regimen in PTPs
Time Frame: For PTPs: up to 5 years or the time it takes to achieve 100 exposure days (EDs).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Bleeds/Year/Subject
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
Number analyzed (Participants) | 49 | 0
Bleeds/Year/Subject
  7-Day Regimen | 0.57 (1.192) |
  (10 or 14)-Day Regimen | 1.05 (2.022) |

ADVERSE EVENTS:
Time Frame: For PTPs: up to 5 years or the time it took to achieve 100 exposure days (EDs). For PUPs: up to 3 years or the time it took to achieve 50 EDs.
Description: Safety Population was used.
Arm/Group | CSL654 (PTPs) | CSL654 (PUPs)
All-Cause Mortality (participants affected / at risk) | 1/83 | 0/12
Serious Adverse Events (participants affected / at risk) | 17/83 | 5/12
Other Adverse Events (participants affected / at risk) | 69/83 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL654 (PTPs) (N=83) | CSL654 (PUPs) (N=12)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0)
Anti factor IX antibody increased (Investigations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abscess Jaw (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL654 (PTPs) (N=83) | CSL654 (PUPs) (N=12)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (3)
Selective IgA immunodeficiency (Immune system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 15 (24) | 6 (9)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (12) | 2 (6)
Laceration (Injury, poisoning and procedural complications) | 6 (7) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 4 (6)
Head injury (Injury, poisoning and procedural complications) | 3 (4) | 3 (5)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Factor VII deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 11 (21) | 0 (0)
Tongue biting (Nervous system disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 10 (12) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (3)
Teething (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (4)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (35) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (25) | 3 (14)
Gastroenteritis (Infections and infestations) | 10 (10) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 1 (2)
Sinusitis (Infections and infestations) | 5 (6) | 0 (0)
Tonsillitis (Infections and infestations) | 5 (8) | 0 (0)
Bronchitis (Infections and infestations) | 4 (8) | 2 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 3 (7)
Ear infection (Infections and infestations) | 3 (3) | 1 (2)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (3)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (2)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Eyelid boil (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Otitis media viral (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02053792/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02053792/SAP_001.pdf